

**Project Title:** EDUCAT: An Assistive Powered Wheelchair. Stage 2. Powered Wheelchair User Evaluation of an Obstacle Alerting System.

NCT Number: NCT05292690

**Document Date: 29/06/2020** 



IRAS ID: 257062

Site Name:

Participant Identification Number for this trial:

## **CONSENT TO USE IMAGES FORM**

Title of Project: EDUCAT An Assistive Powered Wheelchair – Stage 2: User Evaluation of an Obstacle Alerting System

Name of Researcher:

As part of this research study, we would like to take some photographs and/or video clips for data analysis and evaluation.

- These images will be held securely and may be retained in both paper and electronic formats, as part of the record of this evaluation and any associated reports, in accordance with the General Data Protection Regulation (GDPR 2018).
- This consent form limits the use of your images to the purposes that you select below.
- Refusal to give your consent for any of the listed purposes will not affect your participation in this study.
- You may withdraw your consent at any time, by contacting (Insert name of PI and/or local site researcher) contact details below.

Please add your initials into the appropriate box to indicate your choice.

| | | YES | NO |
|---|---|---|---|
| 1. | Would you be happy to consent to photographic and video images | | |
| | being taken for use within this research study? | | |
| 2. | Do you want these images to be anonymised? i.e. face pixelated | | |
| 3. | Would you be happy for these images to be used within associated | | |
| | professional reports, conference presentations and potential | | |
| | publications? | | |
| 4. | Would you be happy to consent to images being used to promote this | | |
| | research study via websites and social media? For example, the | | |
| | EDUCAT website and (insert organisational name). | | |
| | I understand that (organisational name) can have no control over the | | |
| | downloading and use of any images used on public websites. | | |
| 5. | Would you be happy to consent to images being used for promotional | | |
| | purposes by the EDUCAT partner institutions? | | |
| 6. | I have read the above statements and I consent to my images being used for the purposes identified as indicated in the above list. | | |



| Name of Participant | Date | Signature |
|---|---|---|
| Name of Person taking consent | Date | Signature |
| Insert local site contact de | etails – Name of PI and/or | researcher & contact details |
| NB. Original copy for site | filenotes and one copy for | participant. |